CLINICAL TRIAL: NCT04565899
Title: Implementation Intervention to Improve Care for Unhealthy Alcohol Use (CDA 20-057)
Brief Title: Improving Care for Unhealthy Alcohol Use in Primary Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 21-001; K2HX003087 (Other: Department of Veterans Affairs)
Record Dates: First submitted 2020-09-17; First posted 2020-09-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Drinking; Alcohol Use Disorder
Keywords: Unhealthy alcohol use; Alcohol misuse; Alcohol use disorder; Alcohol abuse; Alcohol dependence; Binge drinking; alcohol drinking
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Binge Drinking

STUDY DESIGN:
Intervention Model Description: Pilot trial of an implementation strategy within one primary care clinic where all providers will be invited to participate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Practice facilitation implementation intervention (Experimental): 6 months during which practice facilitation is implemented to support the primary care clinic in improving routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs.
  Interventions: Other: Practice facilitation implementation intervention

INTERVENTIONS:
Other: Practice facilitation implementation intervention — 6 months during which practice facilitation is implemented to support the primary care clinic in improving routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs.

SUMMARY:
In order to improve the quality of alcohol-related care for those with unhealthy alcohol use, the current research will use an evidence-based implementation strategy, practice facilitation, at one VA primary care site to pilot test whether practice facilitation has the potential to improve the quality of primary care-based alcohol-related care . It is hypothesized that primary care providers who take part in the practice facilitation intervention will provide higher quality substance use care to Veterans with unhealthy alcohol use compared to care pre-practice facilitation (e.g., administer evidence-based brief counseling interventions at higher rates, prescribe alcohol use disorder pharmacotherapy at higher rates, increase referrals to specialty substance use disorder clinics).

DETAILED DESCRIPTION:
Alcohol use is a significant risk factor of disability and death for U.S. adults and one out of every six Veterans seen in primary care report unhealthy alcohol use. Based on substantial evidence from randomized controlled trials and the U.S. Preventive Services Task Force, VA/DoD clinical guidelines stipulate that all Veterans screening positive for unhealthy alcohol use should receive evidence-based alcohol care in primary care, including brief counseling interventions (BI) and additional treatment (e.g., pharmacotherapy) for those with alcohol use disorders (AUD). The VA was a pioneer in implementing alcohol screening and BI in primary care, yet substantial implementation gaps remain. In order to improve the quality and fidelity of alcohol-related care, the current research proposes to use an evidence-based implementation strategy, practice facilitation, at one VA to pilot test whether practice facilitation has the potential to improve quality of primary care-based alcohol-related care.

The project will first conduct qualitative interviews assessing Veteran and clinical stakeholders to understand barriers and facilitators to high-quality alcohol care. Results from qualitative interviews will be used to refine and hone the practice facilitation intervention. Clinical stakeholders will then be recruited to participate in focus groups in order to evaluate the acceptability and feasibility of the proposed practice facilitation intervention prior to testing it. Last, a pilot test of the practice facilitation intervention will be conducted within one VA primary care clinic to understand whether practice facilitation improves the quality of primary care-based alcohol-related care.

ELIGIBILITY:
Inclusion Criteria:

Veteran patients:

* Veteran presenting for care at VA primary care site during pilot testing of the practice facilitation intervention, AND
* Age 18 years and older.

Primary care providers:

* Primary care staff who screen for unhealthy alcohol use and providers who practice at the primary care clinic at least 1 day per week.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Reach of alcohol-related care via electronic health record change | 3- and 6-months post implementation intervention
  Reach outcomes will be expressed as a rate, with the denominator (for all outcomes) defined as all Veterans with a visit to the primary care site during active implementation of the practice facilitation pilot test. The numerator for each Reach outcome is as follows: the number of Veterans who screened positive for unhealthy alcohol use (AUDIT-C >= 5) AND had any documented brief intervention, specialty addictions treatment (inpatient and outpatient clinic visits for substance use disorder treatment encounters with an accompanying AUD diagnosis), or pharmacotherapy for AUD (any filled prescription for FDA-approved medications: acamprosate, disulfiram, or oral/injectable naltrexone) in the 30 days following a positive screen. Rates at the start of active implementation and at 3- and 6-months post Active Implementation will be calculated to examine change in Reach outcomes over time.
Adoption of alcohol-related care via electronic health record change | 3- and 6-months post implementation intervention
  Adoption outcomes will be identified as the percentage of providers from the primary care clinic who deliver alcohol-related care when a Veteran screens positive for unhealthy alcohol use (e.g., delivery of brief interventions, consults to specialty addictions treatment, providing pharmacotherapy for AUDs). Rates of alcohol-related care at the start of active implementation and at 3- and 6-months post active implementation will be used to measure whether adoption rates of alcohol-related care increased over time.
Adoption of alcohol related care via self-report change | 3- and 6-months post implementation intervention
  Brief self-report questions to determine whether providers have adopted the suggested evidence-based components of alcohol-related care (e.g., shared decision making, patient-centered discussions, setting goals with patients) will be administered at the start of the active implementation phase, at the end of the active implementation phase, and 3- and 6-months post practice facilitation.
Maintenance of alcohol-related care via electronic health record | 12-months post implementation intervention
  Reach and Adoption outcomes using electronic health record data will be assessed again at 12-months post active implementation to examine whether high-quality alcohol care was sustained after practice facilitation.

SECONDARY OUTCOMES:
Clinical Effectiveness via electronic health record | 12-months post implementation intervention
  Examine whether Veterans' with an encounter in primary care during active implementation reduced their drinking 12-months post Active Implementation using AUDIT-C scores.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L. Bachrach, PhD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Emily C. Williams, PhD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying publications resulting from the proposed research may be shared.
Time Frame: After Oct. 1, 2025
Access Criteria: A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. The limited dataset will be made available following written (email) request to the PI.

REFERENCES:
- [Derived] Bachrach RL, Chinman M, Rodriguez KL, Mor MK, Kraemer KL, Garfunkel CE, Williams EC. Using practice facilitation to improve alcohol-related care in primary care: a mixed-methods pilot study protocol. Addict Sci Clin Pract. 2022 Mar 14;17(1):19. doi: 10.1186/s13722-022-00300-x. PMID 35287714

DOCUMENTS (1):
  • Informed Consent Form (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT04565899/ICF_000.pdf